CLINICAL TRIAL: NCT04785339
Title: Latinx Acculturative Stress Intervention Development and Implementation (REACH Equity CDA)
Brief Title: Acculturative Stress Intervention (REACH Equity CDA)
Acronym: REACH Equity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving institution.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00105969
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2021-11

CONDITIONS: Acculturative Stress
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: * Aim 1: Co-develop an acculturation stress intervention for adult Latinx immigrants to decrease stress, increase resilience, and prevent declines in mental and physical health.
  * Aim 2: Examine the preliminary clinical impact, feasibility, and acceptability of a group acculturative stress in Latinx immigrants and collect information to inform subsequent implementation.
  Aim 2a: Conduct pilot testing of the group intervention in Latinx immigrant participants (N=24-30) to evaluate its preliminary clinical impact from baseline to post-assessment on stress, resilience, and health outcomes (e.g., depression, anxiety, self-rated health).
  o Aim 2b: Characterize the inner and outer context, facilitators, barriers, intent to adopt, and resources across the Duke University Health System through multiple stakeholder interviews with providers and administrators (n=8-10).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one-arm, pre-post design (Experimental): This study will test an intervention in adult Latinx immigrants. There will be no control condition or other comparators. One condition will only provide data at pre (baseline) and post. The only comparison will be across time, but not across conditions as this will be the only condition and all participants will receive the same intervention.
  Interventions: Behavioral: intervention in adult Latinx immigrants

INTERVENTIONS:
Behavioral: intervention in adult Latinx immigrants — Participants will complete self-report outcome measures at pre (baseline) and post, and they will receive the intervention in-between these assessments. Thus, the time frame for data collection is 10 weeks.

SUMMARY:
The overarching aim of the study is to garner empirical support for intervention components that can reduce acculturative stress in Latinx immigrants. Informed by our review of the literature and our prior research, we hypothesize that we can target the following mechanisms in a modularized group intervention format, as detailed below. These are preliminary areas targeted by the intervention, but may be updated based on feedback from the Community Advisory Board, Community Consultation Studio, and Duke Health key informants.

DETAILED DESCRIPTION:
As health disparities widen for Latinx immigrants, there is an urgent unmet public health need to develop an evidence-based interventions reducing stress experienced by this population that can be easily scalable across diverse clinical settings and geographically distinct immigrant communities. Thus, the purpose of this study is to develop and pilot test a novel group acculturative stress intervention for Latinx immigrants.

Study activities Aim 1: Co-develop an acculturation stress intervention for adult Latinx immigrants to decrease stress, increase resilience, and prevent declines in mental and physical health.

Aim 2: Examine the preliminary clinical impact, feasibility, and acceptability of a group acculturative stress in Latinx immigrants and collect information to inform subsequent implementation.

Aim 2a: Conduct pilot testing of the group intervention in Latinx immigrant participants (N=24-30)to evaluate its preliminary clinical impact from baseline to post-assessment on stress, resilience, and health outcomes (e.g., depression, anxiety, self-rated health).

Aim 2b: Characterize the inner and outer context, facilitators, barriers, intent to adopt, and resources across the Duke University Health System through multiple stakeholder interviews with providers and administrators (n=8-10).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old,
* Latinx/Hispanic Self identifying
* Immigrant (born outside of the US)

Exclusion Criteria:

* Active suicidal ideation (i.e., imminent SI in the last 12 months AND ≥1 suicide attempts in the last 10 years)
* Unmanaged severe mental illness (i.e., psychotic disorder, manic symptoms, eating disorder, substance use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Acculturative Stress as measured by the Hispanic Stress Inventory-2 | 10 weeks
  Hispanic Stress Inventory-2 is 24 item questionnaire asking about stress on a scale of 1 to 5, where 1 is not stressed and 5 is very stressed".
Perceived Stress as measured by the Perceived Stress Scale | 10 weeks
  The Perceived Stress scale is a 23-item questionnaire asking about stress on a scale of 1 to 5, where 1 is not stressed and 5 is extremely stressed.
Dispositional resilience as measured by the Resiliency Scale | 10 weeks
  Resilience scale is a 25-item questionnaire asking resilience on a scale of 1 to 7, where 1 is disagree and 7 is strongly agree.
Coping strategies as measured by the Brief COPE Scale | 10 weeks
  Brief COPE Scale is a 24-item questionnaire asking coping on a scale of 1 to 4, where is not at all and 4 is a lot.
Ethnic Identity as measured by the Multigroup Ethnic Identity Measure | 10 weeks
  MEI is a 12-item questionnaire asking about Hispanic identity on a scale of 1 to 7, where 1 is strongly disagree and 7 is strongly agree.
Familism as measured by Familism Scale. | 10 weeks
  Familism Scale is a 15 -item questionnaire asking about family welfare concern on a scale of 1 to 6, where 1 is strongly disagree and 6 is don't know.
Social Support as measured by Social Support Questionnaire | 10 weeks
  Social Support Questionnaire is 16-item questionnaire asking about social support on a scale of 1 to 5, where 1 is Never and 5 is always.

SECONDARY OUTCOMES:
Anxiety symptoms as measured by GAD-7 | 10 weeks
  Generalized Anxiety Disorder survey is a 7-item questionnaire asking problems anxiety on a scale 1 to 4, where 1 is not at all and 4 is Nearly every day.
Depression symptoms as measured by PHQ-9 | 10 weeks
  PHQ-9 is a self-reported patient health questionnaire survey is a 9 - item on a scale of 1 to 4, where 1 is Not at all and 4 is Nearly every day.
Sleep Disturbance as measured by Sleep Disturbance | 10 weeks
  Sleep disturbance is a self-reported 4 questionnaire survey on a scale of 1 to 5, where 1 is very poor and 5 is very good.
Drug Use as measured by Drug Abuse screening Test (DAST) | 10 weeks
  Drug use is asking the use of prescribed, over the counter in excess of direction and any nonmedical use of drugs on a scale of yes and no.
Self-reported Physical Health as measured by Physical activity. | 10 weeks
  physical activity is a self-reported 2 questionnaire on a scale of 0 to 7.
Self-reported Physical Health as measured by Short Form Health Survey | 10 weeks.
  Short Form Health Survey is a 19-item self reported questionnaire on a scale of 1 to 5, where 1 is poor and 5 is Excellent.
Self-reported Physical Health as measured by Self-Rated Health | 10 weeks
  Self- Rated Health is a 7-item questionnaire on a scale of 1 to 5, where 1 is Excellent and 5 is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Nagy, Ph.D., Principal Investigator — Duke Health

IPD SHARING:
Plan to Share IPD: No